CLINICAL TRIAL: NCT06710210
Title: Hybrid Percutaneous Coronary Intervention Combining a Bioresorbable Scaffold With Drug-coated Balloons Versus a Conventional Drug-eluting Stent-based Strategy in Patients With Long and Diffuse Coronary Artery Disease: the BIOHYBRID Randomized Pilot Trial
Brief Title: Hybrid Percutaneous Coronary Intervention Combining a Bioresorbable Scaffold With Drug-coated Balloons Versus a Conventional Drug-eluting Stent-based Strategy in Patients With Long and Diffuse Coronary Artery Disease
Acronym: BIOHYBRID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Clinical Trials Unit Bern (CTU) (Unknown)
Responsible Party: Principal Investigator, IGLESIAS Juan Fernando, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0000
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Diffuse Coronary Artery Disease; Percutaneous Coronary Intervention (PCI)
Keywords: Diffuse/long coronary artery disease; Percutaneous coronary intervention; Drug-eluting stents; Drug-coated balloons; Bioresorbable scaffold
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid PCI strategy (Experimental): Hybrid percutaneous coronary intervention with a bioresorbable scaffold and drug-coated balloon(s)
  Interventions: Device: PCI with a bioresorbable scaffold and drug-coated balloon(s)
- Conventional PCI strategy (Active Comparator): Percutaneous coronary intervention with drug-eluting stent(s)
  Interventions: Device: PCI with drug-eluting stent(s)

INTERVENTIONS:
Device: PCI with a bioresorbable scaffold and drug-coated balloon(s) — Hybrid PCI combining a magnesium-based sirolimus-eluting bioresorbable scaffold (Freesolve, Biotronik AG, Switzerland) and ≥1 paclitaxel-eluting drug-coated balloon(s) (Pantera Lux, Biotronik AG, Switzerland)
  Arms: Hybrid PCI strategy
Device: PCI with drug-eluting stent(s) — PCI with >1 newer-generation drug-eluting stent (Orsiro Mission, Biotronik AG, Switzerland)
  Arms: Conventional PCI strategy

SUMMARY:
The primary objective of the study is to assess the safety and the efficacy of a hybrid percutaneous coronary intervention (PCI) strategy combining a magnesium-based sirolimus-eluting bioresorbable scaffold (Freesolve, Biotronik AG, Switzerland) and ≥1 paclitaxel-eluting drug-coated balloon(s) (Pantera Lux, Biotronik AG, Switzerland) compared to a conventional DES-based PCI approach using >1 newer-generation drug-eluting stents (Orsiro Mission, Biotronik AG, Switzerland) for the treatment of patients with long and/or diffuse coronary artery lesions suitable for PCI with respect to vessel-level absolute change in non-invasive angiography-derived fractional flow reserve (FFRangio, CathWorks, Newport Beach, USA) between post-index PCI and 12-month follow-up.

BIOHYBRID is a coronary revascularization strategy study comparing two contemporary treatment approaches for patients with long and/or diffuse coronary artery lesions undergoing PCI.

The primary hypothesis of the study is that a hybrid PCI strategy using a 'leave nothing behind' or 'metal-free' approach that combines a bioresorbable magnesium scaffold and drug-coated balloons for the treatment of patients with long and/or diffuse coronary artery lesions suitable for PCI is feasible.

The secondary hypothesis is that a hybrid PCI strategy combining a bioresorbable magnesium scaffold and drug-coated balloons is non-inferior to a conventional DES-based PCI approach using one or several DES for the treatment of patients with long and/or diffuse coronary artery lesions suitable for PCI with respect to vessel-level absolute change in FFRangio (CathWorks, Newport Beach, USA) between post-index PCI and at 12 months of follow-up.

DETAILED DESCRIPTION:
1. Newer-generation drug-eluting stents for the treatment of de novo coronary artery disease Among patients with significant coronary artery disease (CAD) undergoing percutaneous coronary intervention (PCI), the use of newer-generation drug-eluting stents (DES) is currently recommended in all patients and lesions subsets. However, despite modern iterations in DES designs including reduced stent strut thickness, improved polymer biocompatibility and/or resorption, and controlled antiproliferative drug release, long-term clinical outcomes after PCI in patients with CAD are not further improving. In a patient-level pooled analysis of 19 prospective randomized controlled trials including 25,032 patients undergoing PCI, of which 13,380 underwent PCI with second-generation DES, very-late stent-related events occurred between 1 and 5 years after PCI at a rate of ∼2%/year with all stent types, with no plateau evident, highlighting the need for new approaches to improve long-term outcomes after PCI. Among potential responsible mechanisms, the persistence of a metallic stent platform and a permanent polymer coating prevents vasomotion and positive coronary artery remodelling, and triggers inflammation, neoatherosclerosis and stent fracture which may lead to in-stent restenosis or very late stent thrombosis. These findings highlight the need for novel iterations of DES technologies and innovative PCI approaches to overcome the persisting limitations of current generation DES for the treatment of patients with CAD.
2. Percutaneous coronary intervention for de novo long and/or diffuse coronary artery disease Patients with de novo long and/or diffuse CAD undergoing PCI represent a particularly challenging clinical subset and remain an unmet clinical need for the interventional community. De novo long and/or diffuse coronary lesions are found in 20% of patients undergoing PCI and newer-generation DES implantation in patients with long and/or diffuse CAD is associated with an increased risk of stent failure at long-term follow-up. In a patient-level pooled analysis from the GRAND-DES registry including 9,217 patients from five Korean multicenter DES registries, 1,182 patients (13%) underwent long stenting (>40 mm) with contemporary second-generation DES. At a median follow-up duration of 2 years, long stenting was associated with significantly higher rates of target lesion failure (TLF), defined as the composite of cardiac death, target vessel myocardial infarction, or clinically indicated target lesion revascularization (8.1% vs. 4.5%, IPTW adjusted HR 1.88, 95% CI: 1.67-2.13; p<0.001), and definite or probable stent thrombosis (1.0% vs. 0.4%, IPTW adjusted HR 2.20, 95% CI: 1.51-3.20; p<0.001) compared with shorter stenting (≤40 mm). Target vessel failure (TVF), defined as the composite of cardiac death, target vessel myocardial infarction, or clinically indicated target vessel revascularization, at 2 years were 10.8% vs. 6.0% in the long and short stenting groups, respectively. Diffuse long lesions commonly require stenting with long (≥ 60 mm) overlapping DES, which is a known predictor of adverse events such as in-stent restenosis or stent thrombosis. Furthermore, particularly for young patients with long and/or diffuse coronary lesions, the 'full metal jacket' with metallic DESs may preclude the possibility of future surgical revascularization options.
3. Hybrid percutaneous coronary intervention for de novo long and/or diffuse coronary artery disease Given the recent data supporting the safety and efficacy of a drug-coated balloon (DCB)-only strategy in patients with small vessel CAD in addition to the natural step-down of vessel diameter in de novo long and/or diffuse coronary lesions, a hybrid PCI approach combining a newer-generation DES (implanted at the larger, more proximal, segment of the lesion) and a DCB (located at the smaller, more distal segment of the lesion) has been recently proposed as a potential alternative treatment strategy for patients with de novo long and/or diffuse coronary artery disease. Hybrid PCI using a single DES combined with DCB instead of several overlapping DES may reduce total stent length, thus minimizing the risk of long-term stent failure. In the prospective, multicenter, observational, non-randomized HYPER study including 106 consecutive patients with de novo diffuse CAD undergoing PCI with a hybrid approach, consisting in the combined use of DES and DCB in contiguous coronary segments, procedural success was 96.2%, and the primary device-oriented composite endpoint (DOCE) of cardiac death, target vessel myocardial infarction and ischemia-driven target lesion revascularization at one year of follow-up was 3.7%, with all the adverse events caused by ischemia-driven target lesion revascularization. Similarly, a previous retrospective study demonstrated that a DCB-only strategy or in combination with DES (hybrid approach) in the treatment of de-novo diffuse CAD (>25 mm), had comparable rates of major adverse cardiovascular events (20.8% vs. 22.7%; p=0.74) and target lesion revascularization (9.6% vs. 9.3%, p=0.84), respectively at 2 years follow up. However, the long-term results of a hybrid PCI strategy combining DES with DCB remain limited by the persisting high rates of stent-related adverse outcomes associated with the use of permanent metallic DES.
4. Bioresorbable scaffolds for the treatment of coronary artery disease Bioresorbable scaffolds (BRS) were developed to overcome the persisting limitations of contemporary DES, enabling vessel restoration and reducing long term risk of device failure after PCI. BRS are hypothesized to provide a temporary drug-eluting scaffold, which supports the vessel after implantation, thus limiting acute recoil and negative remodeling, and enabling a natural biologic reconstruction of the arterial wall and restoration of the vascular function once the scaffold is resorbed.

   Freesolve (Biotronik AG, Bülach, Switzerland) is a third-generation magnesium-based sirolimus-eluting bioresorbable scaffold that has obtained CE mark for coronary use in 2024. This bioresorbable scaffold is built with a refined magnesium alloy and enhances some scaffold properties, such as radial strength, scaffolding time and marker visibility, broadens the size range and reduces crossing profile and strut thickness with the aim to improve device-related clinical outcomes. In the BIOMAG-I first-in-man study that included 116 patients with 117 coronary artery lesions, in-scaffold late lumen loss was 0.21+/- 0.31 mm at 6 months of follow-up. Intravascular ultrasound assessment showed preservation of the scaffold area (mean 7.59 mm2 [SD 2.21] post-procedure vs 6.96 mm2 [SD 2.48]) at six months) with a low mean neointimal area (0.02 mm2 [SD 0.10]). Optical coherence tomography revealed that struts were embedded in the vessel wall and were already hardly discernible at six months. Target lesion failure occurred in one (0.9%) patient; a clinically driven target lesion revascularization was performed on post-procedure day 166. No definite or probable scaffold thrombosis or myocardial infarction was observed. These findings demontrate that the implantation of Freesolve bioresorbable scaffold (Biotronik AG, Bülach, Switzerland) in de novo coronary lesions is associated with favorable safety and performance outcomes, comparable to contemporary drug-eluting stents. At 12 months of follow-up, after completion of resorption, in-scaffold late lumen loss was 0.24±0.36 mm (median 0.19, interquartile range 0.06-0.36). The minimum lumen area was 4.95±2.24 mm² by intravascular ultrasound and 4.68±2.32 mm² by optical coherence tomography. Three target lesion failures were reported (2.6%, 95% confidence interval: 0.9-7.9), all clinically driven target lesion revascularisations. Cardiac death, target vessel myocardial infarction and definite or probable scaffold thrombosis were absent. These results confirm that this third-generation bioresorbable magnesium scaffold is clinically safe and effective, making it a possible alternative to DES. Potential factors contributing to this difference in clinical outcomes compared to other available bioresorbable scaffolds, include different scaffold design and materials, reduced thrombogenicity, as shown in preclinical animal models shorter resorption time, and the BIOlute active coating as that is also used in the Orsiro (Biotronik AG, Bülach, Switzerland) DES that has demonstrated consistently low rates of target lesion failure in several randomized clinical trials.

   With the positive data emerging, a hybrid 'leaving nothing behind' approach combining a BRS with a DCB in de novo long/diffuse coronary artery disease represents a novel promising treatment strategy that may provide additional clinical benefits compared with a hybrid PCI approach combining a DES and a DCB. However, randomized data are currently limited. In a small retrospective study including 42 consecutive patients with diffuse de novo or in-stent restenosis treated with a polymeric-based BRS (ABSORB, Abbott Vascular, USA) implantation (larger proximal segment) and DCB inflation (smaller distal segment or bifurcation side branch), procedural success was obtained in all patients, but three (7.3%) patients required bail-out scaffolding for DCB-related dissections. At a median follow-up of 12 months, there were no cases of cardiac death, target vessel myocardial infarction, or BRS/DCB segment thrombosis. Ischemia-driven target lesion revascularization occurred in two (4.7%) BRS-treated segments. These findings suggest that a hybrid strategy using BRS and DCB in different segments in patients with long diffuse CAD is feasible and associated with encouraging clinical outcomes.

   With increasingly higher rates of diffuse coronary lesions to be treated by means of PCI, and still suboptimal long-term results using the current DES, the need for a new approach to treat these lesions represents an unmet clinical need. Freesolve (Biotronik AG, Bülach, Switzerland) bioresorbable scaffold, with a 12-month resorption time, allows for a long-term metal-free vessel, while at the same time providing the temporary scaffolding benefits. Recent studies demonstrate compelling safety data, low TLF rates even in the long-term, and low rates of scaffold thrombosis even in more complex patients.
5. Coronary physiology assessment following percutaneous coronary intervention Intracoronary physiological assessment is acknowledged as a valuable strategy to identify the presence of flow-limiting epicardial stenoses in patients planned for PCI. Numerous large-scale, prospective, multicenter, randomized outcome trials have demonstrated improved clinical outcomes when measuring fractional flow reserve (FFR) with a coronary pressure wire to guide decision-making regarding coronary revascularization in the cardiac catheterization laboratory. However, PCI does not guarantee optimal myocardial revascularization, i.e., restoration of normal epicardial conductance, and recent studies have shown that residual pressure gradients remain in 10-36% of cases despite angiographically successful PCI. During the last years, coronary physiology assessment following PCI has emerged as a valuable tool to assess and potentially optimize the results of percutaneous coronary revascularization. Post-PCI intracoronary pressure measurements can identify residual flow-limiting disease, differentiate residual focal lesions from diffuse disease and provide prognostic information. In patient-level meta-analysis of 28 studies from 17 cohorts including a total of 5,277 patients with 5,869 vessels who underwent FFR measurement after DES implantation lower post-PCI FFR significantly increased the risk of target vessel failure (TVF) (adjusted hazard ratio [HR] per 0.01 FFR decrease, 1.04; 95% CI, 1.02-1.05; p<0.001). The risk of cardiac death or myocardial infarction also increased inversely with post-PCI FFR (adjusted HR, 1.03; 95% CI, 1.00-1.07, p=0.049). Whereas a higher post-PCI FFR is associated with a lower incidence of adverse clinical outcomes, the cut-off point for an optimal PCI result is still debated. In a systematic review and meta-analysis of 7,470 patients from 105 studies, post-PCI FFR ≥0.90 has been associated with a significantly lower risk of repeat PCI (odds ratio, 0.43; 95% CI, 0.34-0.56; p<0.0001) and major adverse cardiac events (odds ratio, 0.71; 95% CI, 0.59-0.85, p=0.0003) (X).

An important aspect of the previous evidence is that the stent length was relatively short, averaging <20 mm. A recent study demonstrates that this did not translate to patients with diffuse long segment coronary artery lesions requiring long (30-49 mm) or ultralong DES (≥50 mm). In this single-centre prospective study including 74 patients who received long or ultra-long DES, FFR >0.90 immediately after PCI was achieved only in 28.4% (21/74) of patients, of whom only two had received ultralong DES. At 9-month follow-up, 61 patients had FFR measured; 23% of patients had an FFR >0.90, restenosis rate was 15.1% by functional assessment, and target lesion revascularization occurred in 8.1% of patients. The rate of patients achieving FFR >0.90 immediately after PCI and at 9-month follow-up is considerably lower than that reported in the previous studies on shorter stents, suggesting that it is more challenging to achieve satisfactory post-PCI FFR values in patients treated with long or ultra-long DES. One possible mechanism is that patients requiring ultralong stents have a substantial burden of residual diffuse disease. Reduced vascular compliance in long DES is another mechanism for a persistent post-PCI FFR gradient. Healthy coronary vessels and the microcirculation are able to regulate coronary flow even in the presence of atheroma, aiming to balance the coronary flow with myocardial oxygen requirements. Endothelial dysfunction is an accepted phenomenon secondary to mechanical injury of the vessel immediately after stent deployment. Therefore, it is expected that longer stents will cause a larger area of damage, augmenting the process of vascular dysfunction. This leads to a reduction in the endothelial release of vasoactive substances in the stented segment of a long DES. Normal vessel vasomotion is further limited by the larger metallic frame of a long DES producing a greater radial force resistive to changes in vessel diameter. These mechanisms provide a further explanation for lower post-PCI FFR values in long DES and serve as a background to investigate the potential role of a completely 'leave nothing behind' PCI strategy combining bioresorbable scaffolds and drug-coated balloons for the treatment of patients with long/diffuse coronary artery disease.

Measuring FFR with a pressure wire remains underutilized because of the invasiveness of guide wire placement or the need for a hyperemic stimulus. Over recent years, several functional coronary angiography technologies deriving similar information than invasive FFR from an invasive coronary angiogram or non-invasive computed tomography coronary angiography have emerged as a promising non-invasive alternative to wire-based FFR measurement with the objective to streamline coronary physiology assessment in daily practice work-flow. Nowadays, several non-invasive FFR-equivalent modalities derived from invasive coronary angiograms and supported by prospective validation studies are commercially available. The FFRangio system (CathWorks, Newport Beach, USA) is a novel non-invasive angiography-derived coronary physiology index measuring FFR without a coronary pressure wire or hyperemic agent that combines artificial intelligence and advanced computational science to obtain physiologic information from routine angiograms to inform treatment decisions. The FFRangio concept relies on creating a 3-dimensional (3D) reconstruction of the coronary arterial system and estimating the resistance and flow across a coronary stenosis. In the FFRangio Accuracy versus Standard FFR (FAST-FFR) prospective study that included 301 subjects and 319 vessels, FFRangio measured from the coronary angiogram alone has a high sensitivity, specificity, and accuracy compared with pressure wire-derived FFR. The per-vessel sensitivity and specificity were 94% (95% CI, 88% to 97%) and 91% (86% to 95%), respectively, both of which exceeded the prespecified performance goals. The diagnostic accuracy of FFRangio was 92% overall and remained high when only considering FFR values between 0.75 to 0.85 (87%). FFRangio values correlated well with FFR measurements (r=0.80, P<0.001) and the Bland-Altman 95% confidence limits were between -0.14 and 0.12. The device success rate for FFRangio was 99%. In a recent pooled analysis of 5 prospective cohort studies including 700 lesions from 588 patients, FFRangio showed excellent diagnostic performance, which was robust and consistent across all patient and lesion subgroups. When using a binary cutoff FFR value of 0.80, FFRangio showed a sensitivity of 91%, a specificity of 94%, and a diagnostic accuracy of 93%. The mean difference between FFR and FFRangio was 0.00 ± 0.12. The correlation coefficient between FFR and FFRangio was 0.83 (p<0.001). The C-statistic for FFRangio was 0.95 (p<0.001). The accuracy of FFRangio was consistent across all subgroups examined. Accordingly, FFRangio has the promise to substantially increase physiological coronary lesion assessment in the catheterization laboratory, thereby potentially leading to improved patient outcomes. These robust data support the use of FFRangio derived from coronary angiogram as a valid non-invasive alternative to invasive wire-based FFR to assess coronary physiology after PCI without manipulating the coronary artery with its inherent risk of complications and the need for a hyperemic stimulus.

ELIGIBILITY:
Inclusion criteria:

* Clinical inclusion criteria

  1. Participant is ≥18 years.
  2. Participant has provided written informed consent as approved by the independent Ethical Committee (EC) or Institutional Review Board (IRB) of the respective participating centre prior to any study-related procedure.
  3. Participant is eligible for PCI according to the ESC guidelines (4, 5) .
  4. Participant is hemodynamically stable.
  5. Participant with chronic coronary syndrome (CCS) or acute coronary syndrome (ACS): unstable angina, non-ST-segment elevation myocardial infarction (NSTEMI), or stabilized ST-segment elevation myocardial infarction (STEMI).

  5a. Participants with STEMI are eligible for the treatment of non-culprit coronary lesions, if participant consent occurs ≥72 hours after successful primary PCI of the culprit STEMI lesion.

  5b. Target lesion(s) to be treated are not located in the STEMI culprit vessel(s) and are not STEMI culprit lesion(s).

  6. Participant is eligible for dual antiplatelet therapy (DAPT) with aspirin plus either clopidogrel, prasugrel, or ticagrelor for ≥6 months.

  7. Participant is willing to participate and able to comply with the protocol requirements for the duration of the study, including completion of study visits and control coronary angiogram at 12 months.

Angiographic inclusion criteria 8. Target lesion length is >40 mm according to operator visual estimation, which may be assisted by Quantitative Coronary Angiography (QCA), Intravascular Ultrasound (IVUS), or Optical Coherence Tomography (OCT).

9. Target vessel has a maximum reference diameter between 3.0-4.6 mm according to operator visual estimation, which may be assisted by QCA, IVUS, or OCT.

Notes: The proximal segment, which has a larger vessel diameter, will be treated with one Freesolve scaffold, in accordance with the vessel diameter range specified in the IFU. The distal segment, which naturally tapers to a smaller diameter, can be treated with one or more Pantera Lux DCB, in accordance with the vessel diameter range specified in the IFU.

10. Target lesion with a baseline (pre-PCI) Thrombolysis In Myocardial Infarction (TIMI) flow ≥1.

Exclusion criteria:

Clinical exclusion criteria

1. Participant has a known allergy to contrast medium that cannot be adequately premedicated, or any known allergy or intolerance to aspirin, P2Y12 receptor inhibitors (clopidogrel, ticagrelor, or prasugrel), both heparin and bivalirudin, any of the following DES or bioresorbable scaffold component (magnesium, aluminium, tantalum, poly-L-lactide, or sirolimus), or drug-coated balloon component (paclitaxel).
2. Participant with STEMI <72 hours prior to study index procedure. 12a: Participants with hemodynamically stable NSTEMI are eligible for study enrolment.
3. Participant with prior PCI within the target vessel during the last 12 months prior to the study index procedure.
4. Participant is on dialysis or has chronically impaired renal function defined as serum creatinine >2.5 mg/dL or 221 μmol/L.
5. Participant is unable to adhere to DAPT for at least 6 months (e.g. planned surgery, dental surgical procedure, active bleeding disorders, active coagulopathy).
6. Participant is on oral anticoagulation therapy (OAC) prior to index procedure unless DAPT plus OAC (i.e. triple therapy) can be maintained for a minimum of 1 month.
7. Participant with life expectancy <1 year.
8. Participant is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study.
9. Participant is currently participating or planning to participate in another interventional clinical trial, except for observational registries or previous enrolment into the current investigation.
10. Participant unwilling or unable (e.g. physical or cognitive) to comply with study procedures, medication adherence and schedule.
11. Contraindications and limitations of the medical devices as described in the instructions for use.
12. Known or suspected non-compliance, drug or alcohol abuse.
13. Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
14. Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation.

    Angiographic exclusion criteria
15. Target vessel previously treated with a bare-metal stent or a drug-eluting stent and the target lesion is within 5 mm proximal or distal to the previously treated lesion.
16. Target lesion is a chronic total occlusion.
17. Target lesion is located in left main coronary artery, ostial left anterior descending artery, ostial left circumflex artery, or ostial right coronary artery (within 5.0 mm of the vessel origin).
18. Target lesion is located in, or supplied by, an arterial or venous bypass graft.
19. Target lesion with excessive tortuosity proximal to or within the lesion based on operator visual estimation, or heavily calcified target lesion which may be adequately prepared using a non-compliant and/or cutting/scoring balloon.
20. Target lesion requires treatment with a device other than a non-compliant balloon and/or a modified (cutting/scoring) balloon prior to scaffold/stent placement (including but not limited to atherectomy devices, intravascular lithotripsy).
21. Target lesion involves a coronary bifurcation with a side branch with reference vessel diameter ≥2.0 mm that requires a two-device strategy after pre-dilatation.
22. Presence of thrombus in the target vessel.
23. Future planned staged PCI or coronary artery bypass graft surgery after the study PCI procedure.
24. Target with unsuccessful lesion preparation, defined as the absence of residual stenosis ≥30%, TIMI flow grade <3 following complete lesion preparation (6), type C to F coronary artery dissection according to the National Heart, Lung and Blood Institute (NHLBI) classification (7) (Appendix 2) and angiographic complications (e.g. distal embolization, or side branch closure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Vessel-level delta FFRangio values between post-PCI and 12-month follow-up | 12 months
  Vessel-level delta angiography-derived Fractional Flow Reserve values between post-PCI and 12-month follow-up

SECONDARY OUTCOMES:
Vessel-level FFRangio value after index PCI | After index PCI
  Vessel-level angiography-derived fractional flow reserve value after index PCI
Vessel-level FFRangio value at 12-month follow-up | 12 months
  Vessel-level angiography-derived Fractional Flow Reserve value at 12-month follow-up
Rate of target vessel failure | 12 months
  Composite of cardiac death, target vessel myocardial infarction, or clinically indicated target vessel revascularization

OTHER OUTCOMES:
Rate of vessel-oriented composite endpoint (VOCE) | 12 months.
  Composite of vessel-related cardiac death, vessel-related myocardial infarction, or target vessel revascularization
Rate of all-cause death | 12 months
  Cardiac and non-cardiac death
Rate of any myocardial infarction | 12 months
  Periprocedural or spontaneous, Q wave or non-Q wave, myocardial infarction
Rate of any revascularization | 12 months
  PCI or CABG, clinically and not clinically indicated target lesion revascularization, clinically and not clinically indicated target vessel revascularization
Rate of definite and definite/probable device thrombosis | 12 months
  Academic research Consortium definite and definite or probable device thrombosis
Rate of major bleeding | 12 months
  Bleeding Academic research Consortium (BARC) 3 or 5 major bleeding events
Rate of Target Lesion Revascularization | 12 months
  Clinically and not clinically indicated Target Lesion Revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD and relevant documentation will be made available to external investigators not affiliated to the trial who provide a detailed study protocol according to international guidelines and whose proposed use of the data has been approved by the study principal investigator.